CLINICAL TRIAL: NCT04751630
Title: Effects of a Structured Online Therapeutic Exercise Program on Physical Performance in COVID-19 Patients at Discharge Time.
Brief Title: Effects of COVID-19 Hospitalization on Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Doctor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS-21-22
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Physical Disability
MeSH Terms: conditions — COVID-19 | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercise group (Experimental): The study participants corresponding to the Therapeutic Exercise (ET) intervention group will follow the prescriptions given to them by their primary care physician. In addition, and as the main part of the intervention, they will undergo a six-week ET program with two sessions per week, for a total of 12 sessions. Full participation in 10 sessions will be necessary to be included in the ET group during the statistical analysis. Each session will be one hour long. The sessions will be given and supervised by a physiotherapist expert in therapeutic exercise prescription through the online modality.
  Interventions: Other: Therapeutic Exercise
- Control group (No Intervention): Study participants in the control group will follow the prescriptions given to them by their primary care physician and will receive a weekly call to assess their recovery. At the end of the study follow-up, when their participation in the study as a control group ends, participants in this group will be offered to participate in the structured ET program to be carried out by the ET group. The reason for this is to ensure that the entire sample ends up receiving a treatment that, a priori, should improve their functional capacities, thus guaranteeing one of the ethical principles of the research.

INTERVENTIONS:
Other: Therapeutic Exercise — Online and structured exercise therapeutic program based on flexibility, strength, balance and aerobic exercises. The program have been supervised by an expert on the field and it participants will perform it under the supervision of an expert physiotherapist.
  Arms: Therapeutic Exercise group

SUMMARY:
Coronavirus disease (COVID-19) has resulted in millions of hospital admissions. The physical consequences caused by COVID-19 hospitalization could jeopardize the overall health status of patients through a decrease in functional capacity. A therapeutic exercise program may reduce the adverse effects of COVID-19 on functional capacity and thereby improve the overall health status of these patients.

The objectives of this project are 1) to analyze the effect of a therapeutic exercise program in patients who have been hospitalized in Intensive Care Unit (ICU) for COVID-19.

Single-blind randomized clinical trial. 118 patients post-ICU for COVID-19 will be randomized into an intervention group and a control group. The intervention group will perform a therapeutic exercise program for eight weeks in telematic modality. Functional capacity will be analyzed using the grip strength, Short Physical Performance Battery, gait speed, lower extremity strength and the FRAIL scale at baseline, eight and twelve weeks. The main statistical analysis will be a comparison of means for independent samples assessing the effect of the intervention.

Given the high prevalence of patients hospitalized for COVID-19, establishing strategies to minimize the adverse effects of the virus on patients is a must for the healthcare setting. Assessing physical condition after COVID-19 will allow the magnitude of the problem to be established. Physiotherapy, through therapeutic exercise, could improve physical fitness in these patients and thus improve the overall health status after COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Have been diagnosed COVID-19 positive at the time of hospital admission.
* Be able to use an online platform to conduct "meetings" with the healthcare professional or have the necessary personal assistance to do so.
* Be able to read the informed consent form and understand the objectives and conduct of the study.

Exclusion Criteria:

* Diagnosed neurological or psychiatric disease.
* Contraindications to physical exercise.
* Failure to give informed consent for the study.
* Unavailability to perform the ET program twice a week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Upper limb strength change | Change from Baseline upper limb strength at 6 weeks
  handgrip strength test

SECONDARY OUTCOMES:
Physical Performance change | Change from Baseline physical performance at 6 weeks
  Short Physical Performance Battery test
Walking speed change | Change from Baseline walking speed at 6 weeks
  4 meters walking speed
lower limb strength change | Change from Baseline lower limb strength at 6 weeks
  5 times sit and reach test
Fraility change | Change from Baseline fraility at 6 weeks
  FRAIL scale

CONTACTS AND LOCATIONS:
Overall Officials: Albert Pérez-Bellmunt, PhD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Hospital Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided